CLINICAL TRIAL: NCT03310255
Title: Helicobacter Pylori Infection in Renal Transplant Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelmoniem Abdallah Mohamed, Principal Investigator at the department of Tropical medicine and gastroenterology, Assiut University
Other Study IDs: HPRD
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Helicobacter Pylori Infection; Renal Transplant Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: H pylori Faecal Antigen — All patients will be screened for H. pylori using fecal Ag and positive patients will do endoscopy and biopsy.
  Other Names: Endoscopic Biopsy and culture; PCR

SUMMARY:
Upper gastrointestinal (GI) symptoms are frequent in organ transplant recipients. Peptic ulcers and related pathologies such as gastritis and duodenitis are known to occur with increased frequency (20-60%) and severity in renal transplant recipients. The frequency of severe complications is about 10% among transplant recipients and 10% of those might prove fatal As kidney transplant recipients have to take immunosuppressive drugs for a lifetime and because these drugs have many side effects that may not be differentiated from H. pylori infection Thus, in order to reduce the use of medications and subsequently to reduce the drug interactions ,proper detection and management of H pylori infection in those patients is preferred.

DETAILED DESCRIPTION:
The prevalence of HP colonization is about 30% in the United States and other developed countries as opposed to more than 80% in most developing countries.

Essentially, all HP-colonized persons have gastric inflammation, but this condition in itself is asymptomatic.

Upper gastrointestinal (GI) symptoms are frequent in organ transplant recipients. Peptic ulcers and related pathologies such as gastritis and duodenitis are known to occur with increased frequency (20-60%) and severity in renal transplant recipients. The frequency of severe complications is about 10% among transplant recipients and 10% of those might prove fatal.

GI complications might require dose reduction or the discontinuation of some of the immunosuppressive medications, affecting graft survival.

Considering the strong body of evidence supporting causal effects of HP infections on the development of peptic ulcers and gastric malignancies, the argumented rate of gastrointestinal complaints may bebattributed to increased HP infection rate among this population.

Few studies have investigated the prevalence of HP infection; about 30% to 40% of renal transplant recipients shown HP colonization of the stomach There are conflicting data about the prevalence of H pylori infection in renal transplant recipients. Most of these studies used anti HP IgG to diagnose H. pylori infection that lack consistent sensitivity and specificity.

Nasri and his colleagues in 2013 concluded significant positive association of serum H. Pylori IgG antibody titer with renal function in renal transplant patient.

As kidney transplant recipients have to take immunosuppressive drugs for a lifetime and because these drugs have many side effects that may not be differentiated from H. pylori infection Thus, in order to reduce the use of medications and subsequently to reduce the drug interactions ,proper detection and management of H pylori infection in those patients is preferred.

There are few studies have investigated the prevalence of HP infection; about 30% to 40% of renal transplant recipients shown HP colonization of the stomach. There are conflicting data about the prevalence of H pylori infection in renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients in the first 1st. year after kidney transplantation.
* Patients diagnosed to have H.pylori infection by H.pylori fecal Ag will do endoscopy and biopsy.

Exclusion Criteria:

* Patients who had previous upper endoscopy with evidence of gastritis or ulcers
* Age more than 65 years old
* Patients with any contraindications to upper endoscopy.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Post renal transplant patients, and patients proven to be h pylori positive will be subjected to further evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Prevalence of H pylori post Renal Transplant Patients | 1 year
  Percentage of H pylori positive patients in post renal transplant patients
Detection of CagA & VacA Genotypes by PCR: | 1 year
  Amplified DNA will be analyzed by agarose gel electrophoresis. The positive sample will produce bands at DNA fragment 138-bp for CagA, 259/286-bp for VacA S1/S2, 290-bp and 352-bp for m1 & m2, respectively.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Mueilo SH. Gastroduodenal lesions and Helicobacter pylori infection in hemodialysis patients. Saudi Med J. 2004 Aug;25(8):1010-4. PMID 15322589
- [Background] Atherton JC, Cao P, Peek RM Jr, Tummuru MK, Blaser MJ, Cover TL. Mosaicism in vacuolating cytotoxin alleles of Helicobacter pylori. Association of specific vacA types with cytotoxin production and peptic ulceration. J Biol Chem. 1995 Jul 28;270(30):17771-7. doi: 10.1074/jbc.270.30.17771. PMID 7629077
- [Background] Nasri H, Rafieian-Kopaei M. Significant association of serum H. pylori IgG antibody titer with kidney function in renal transplanted patients. J Renal Inj Prev. 2013 Mar 1;2(1):23-5. doi: 10.12861/jrip.2013.08. eCollection 2013. PMID 25340117
- [Background] Khedmat H, Ahmadzad-Asl M, Amini M, Lessan-Pezeshki M, Einollahi B, Pourfarziani V, Naseri MH, Davoudi F. Gastro-duodenal lesions and Helicobacter pylori infection in uremic patients and renal transplant recipients. Transplant Proc. 2007 May;39(4):1003-7. doi: 10.1016/j.transproceed.2007.03.034. PMID 17524875
- [Background] Miftahussurur M, Yamaoka Y. Diagnostic Methods of Helicobacter pylori Infection for Epidemiological Studies: Critical Importance of Indirect Test Validation. Biomed Res Int. 2016;2016:4819423. doi: 10.1155/2016/4819423. Epub 2016 Jan 19. PMID 26904678
- [Background] Wu CY, Kuo KN, Wu MS, Chen YJ, Wang CB, Lin JT. Early Helicobacter pylori eradication decreases risk of gastric cancer in patients with peptic ulcer disease. Gastroenterology. 2009 Nov;137(5):1641-8.e1-2. doi: 10.1053/j.gastro.2009.07.060. Epub 2009 Aug 5. PMID 19664631